CLINICAL TRIAL: NCT01329289
Title: Phase II Study of SOM230 LAR in Combination With Bortezomib and Dexamethasone in Patients With Refractory or Relapsed Multiple Myeloma
Brief Title: SOM230 LAR With Bortezomib and Dexamethasone for Refractory or Relapsed Multiple Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Clinical trial being transferred to Columbia University with the Investigator.
Sponsor: University of Pittsburgh (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-078
Record Dates: First submitted 2011-03-29; First posted 2011-04-05 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — pasireotide; Bortezomib; Dexamethasone; Calcium Dobesilate; dexamethasone 21-phosphate; dexamethasone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SOM230 with Bortezomib and Dexamethasone (Experimental)
  Interventions: Drug: SOM230; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: SOM230 — 60 mg intramuscularly (IM) on day 1 of each 28 day cycle
  Other Names: Pasireotide
Drug: Bortezomib — 1.3 mg/m2 intravenously (IV) on days 1, 4, 8, and 11 of each cycle. Bortezomib will be infused by IV push.
  Other Names: Velcade
Drug: Dexamethasone — 20 mg orally on day of and day after bortezomib (Days 1, 2, 4, 5, 8, 9, 11, 12).
  Other Names: Decadron; Dexasone; Diodex; Hexadrol; Maxidex; dexamethasone sodium phosphate; dexamethasone acetate

SUMMARY:
The purpose of this study is to determine if adding SOM230 LAR to bortezomib and dexamethasone is better than bortezomib and dexamethasone alone and if it should be investigated further.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed symptomatic MM, Salmon-Durie Stage II or III, International Staging System II or III, or fulfill the CRAB criteria (see Appendix A, B). Patients should have previously been treated with at least one cycle of bortezomib, after which the patient has shown progressive or refractory disease. Finally, patients must meet at least one of the following parameters of measurable disease:

  * Bone marrow plasmacytosis with> 10% plasma cells, or sheets of plasma cells, or biopsy proven plasmacytoma which must be obtained within 6 weeks prior to registration.
  * Measurable levels of monoclonal protein (M-protein): ≥ 1 g/dL on serum protein electrophoresis (SPEP) or ≥ 200 mg of monoclonal light chain on a 24 hour urine protein electrophoresis (UPEP) or involved FLC ≥ mg/dL (≥ 100 mg/L) which must be obtained within 4 weeks prior to registration.
  * Serum and urine M-protein levels should be determined by electrophoresis rather than by quantitative immunoglobulin (Ig) measurement. Exceptions are made in cases in which the M-spike value may be deemed to be unreliable ( e.g. co-migrating M-spike). In these cases, quantitative Ig should be used. To assess response and progression, however, SPEP values should only be compared to SPEP values and quantitative Ig values only to quantitative Ig values.
* Patients must have received at least two prior anti-MM treatments. The prior treatments must include at least one IMiD (thalidomide or lenalidomide) and bortezomib. If patients are unable to tolerate thalidomide or lenalidomide they can be included without prior IMiD treatment. Patients may be included if they did not experience grade III neuropathy while on bortezomib. Patients may have previously received autologous or peripheral blood stem cell transplantation.
* Minimum of four weeks since any major surgery, completion of radiation, or completion of all prior systemic anticancer therapy. Exception: e.g. kyphoplasty, vertebroplasty, local radiation therapy for symptomatic bone lesions (e.g., uncontrolled pain or high risk of pathologic fracture).
* Age ≥ 18 years.
* Life expectancy of greater than 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%; see Appendix B).
* Patients must have adequate organ and marrow function as defined below, obtained within 4 weeks prior to registration:

  * Hgb > 9 g/dL (which may be supported by transfusion or growth factors)
  * Absolute neutrophil count > 1000 x 10-9/L
  * Platelets ≥ 50,000 x 10-9/L
  * PT/PTT < 1.5 x upper limits of normal (ULN)
  * Total bilirubin ≤ 1.5 x (ULN)
  * Hepatic:

Serum bilirubin ≤ 1.5 ULN

Aspartate aminotransferase and alanine aminotransferase

* 3 × ULN without liver metastases
* 5 × ULN if documented liver infiltration

  * Renal:

Calculated creatinine clearance ≥40 ml/min according to the formula in Appendix D

* Cholesterol* ≤ 300 mg/dL
* Triglycerides (fasting)* ≤ 2.5 x ULN
* Fasting plasma glucose (FPG)** < 1.5X ULN for FPG or HbA1c ≤ 8% *In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.

At the principle investigator's discretion, non-eligible patients can be re-screened after adequate medical therapy has been instituted.

* Patients must not be pregnant or breast feeding and must have a negative pregnancy test within 14 days of the administration of the first study treatment. Further, all women of childbearing potential and sexually active males must agree to use a medically effective contraception method throughout the treatment period and avoid conception while participating in this study. Women must not be lactating. Post menopausal patients and patients who had a bilateral oophorectomy need not take a pregnancy test.
* Ability to understand and the willingness to sign a written informed consent document. Patient must be informed of the investigational nature of this study.
* Patient should be able to swallow pills

Exclusion Criteria:

* Patients who have had chemotherapy, radiotherapy, or major surgery within 4 weeks prior to entering the study or those who have not recovered from AEs due to chemotherapy, radiotherapy, or major surgery completed more than 4 weeks prior to registration. Exception: local radiation therapy for symptomatic bone lesions (e.g., uncontrolled pain or high risk of pathologic fracture).
* Patients with any of the following cardiac abnormalities:

  * QTcF at screening > 450 msec
  * History of syncope or family history of idiopathic sudden death
  * Sustained or clinically significant cardiac arrhythmias
  * Risk factors for Torsades de Pointes such as hypokalemia, hypomagnesemia, cardiac failure, clinically significant/symptomatic bradycardia, or high-grade AV block
  * Concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes, or Parkinson's disease), HIV, cirrhosis, uncontrolled hypothyroidism or cardiac failure
  * Concomitant medication(s) known to increase the QT interval
* Diabetic patients on antidiabetic medications whose HbA1C > 8%
* Patients currently receiving high dose systemic steroids for treatment of MM, patients without prior bortezomib treatment, patients who received an investigational agent within 5 half lives of the agent.
* Patients who require therapeutic (full) anticoagulation such as full dose low molecular weight heparin or Coumadin with a goal INR of 2-3.
* Patients with known brain metastases (treated or not) will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other AEs.
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to SOM230 LAR and/or bortezomib or other agents used in the study.
* Patients should not receive immunization with attenuated live vaccines during study period or within 1 week of study entry.
* Patients with symptomatic cholelithiasis.
* Patients previously treated with sst or sst analogues.
* Patients with a second malignancy other than squamous/basal cell carcinoma of the skin or in situ carcinoma of the cervix unless the tumor was curatively treated.
* Known HIV infection
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * Severely impaired lung function
  * Any active (acute or chronic) uncontrolled disorders
  * Nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the study therapy
* Women who are pregnant or breast feeding, or women/men able to conceive and unwilling to practice a medically effective method of birth control.
* Inability to comply with study and/or follow-up procedures or history of medical noncompliance.
* Patients who have a serious cardiac condition, such as myocardial infarction within 6 months, unstable angina, sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, history of syncope, family history of idiopathic sudden death, QTc > 450 msec, advanced heart block or heart disease as defined by the New York Heart Association Class III or IV. (See ECG guidelines, Section 8.0).
* Patients with non-secretory MM.
* Patients with prior allogeneic transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Objective tumor response | 2 years
  Responses (CR and PR) and incidence of SD will be tabulated by disease diagnosis. All responses will be reported. Response rate among patients with measurable disease will be summarized by exact binomial confidence intervals.

SECONDARY OUTCOMES:
progression-free survival | 2 years
  The progression free survival function will be estimated by means of the product limit (Kaplan-Meier) esitmator with 95% confidence interval. Median PFS will be estimated from the survival function.
Toxicities associated with this investigational combination | 2 years
  Type, incidence severity (NCI-CTCAE grade), timing, relatedness of AE and laboratory abnormalities will be tabulated, with 95% confidence intervals, as appropriate.
Effects of SOM230 LAR on PI3K/MAPK pathway | 2 years
  Serum bone resorption markers, calcium, MIP-1alpha, TRACP-5b, serum (NTx), and serum C-terminal telopeptide (CTx) will be compared to circulating IGF-1 graphically (by scatterplots) and by Pearson or Spearman correlation coefficients, depending on the graphical assessment.
Effect of bortezomib and SOM230 LAR on RANKL production and OCL formation | 2 years
  Serum bone resorption markers will be measured during pretreatment and on day 1 of each cycle. Their change over time will be characterized by estimates derived from a mixed effects ANOVA model.
IGF-1 inhibition and monitor circulating IGF-1 | 2 years
  To analyze whether bortezomib/SOM230 LAR treatment can restore the balance between OCL and osteoblast activity, bone marrow samples will be obtained before treatment and during treatment (day 11 of cycle 2) for OCL formation assays. Mean change over time will be estimated with 95% confidence intervals, and the null hypothesis of no change tested with a paired-comparison t-test
Overall Survival | 5-10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States